CLINICAL TRIAL: NCT04222283
Title: Switch to Tenofovir Alafenamide (TAF), Emtricitabine (FTC), Bictegravir (BIC)(Biktarvy®) in HIV-1-infected Patients Over 65 Years Old at Risk of Polymedication
Brief Title: Switch to TAF+FTC+BIC in HIV-1-infected Patients Over 65 Years Old at Risk of Polymedication
Acronym: BICOLDER
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut de Médecine et d'Epidémiologie Appliquée - Fondation Internationale Léon M'Ba (Other)
Collaborators: Pierre and Marie Curie University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMEA 057
Record Dates: First submitted 2019-12-05; First posted 2020-01-09 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — bictegravir, emtricitabine, tenofovir alafenamide, drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- open label, multicentric, non randomized (Experimental): one arm study to evaluate the safety and efficacy of switching from ritonavir- or cobicistat- booster containing regimens to a fixed-dose combination (FDC) of tenofovir alafenamide (TAF), emtricitabine (FTC) and bictegravir (BIC) in over 65 years old HIV-1-infected patients with virological suppression. Polymedications and drug-drug interactions will be analysed.
  Interventions: Drug: BIKTARVY 50Mg-200Mg-25Mg Tablet

INTERVENTIONS:
Drug: BIKTARVY 50Mg-200Mg-25Mg Tablet — At BSL all the participants will be switched from a booster containing regimen (ritonavir or cobicistat) to TAF/FTC/BIC (BIKTARVY).

SUMMARY:
Patients infected and living with HIV are getting older and have more and more non-HIV co-morbidities. These expose them to polypharmacy that increases the risk of pharmacological interaction. Bictegravir, co-formulated with emtricitabine (FTC) and tenofovir alafenamide (TAF) (BIKTARVY) a new generation integrase inhibitor with a high genetic barrier and had no drug interaction may be a treatment of choice for participant over 65 years old who are HIV infected . BIKTARVY improve adherence and quality of life; and on the other hand it would limit the risks of pharmacological interaction. In addition, the use of TAF reducing the risk of long-term renal toxicity and adverse effects on bone would be of interest in this aging population and more at risk of osteoporosis.

DETAILED DESCRIPTION:
HIV-1-infected patients over 65 years old at risk of polymedication HIV-1-infected adults aged ≥ 65 years who are virologically-suppressed (HIV-1 RNA <50 copies/mL) on a regimen containing a pharmacokinetic enhancer as ritonavir or cobicistat Evaluate the antiviral efficacy of 24 weeks treatment with the fixed dose combination(FDC) of TAF/FTC/BIC

ELIGIBILITY:
Inclusion Criteria:

* HIV-1-infected patient
* Age > 65 years old
* Plasma HIV RNA ≤ 50 copies/mL for ≥ 6 months: one blip between 50 et 200 cp/ml is allowed in the past 6 months before screening.
* Currently receiving an antiretroviral regimen containing a booster, ritonavir or cobicistat
* No resistance mutation to integrase inhibitors on cumulative HIV RNA genotype. The reverse transcriptase resistant mutations M184V plus one TAM are allowed.
* If no genotype is available, DNA genotype will be performed at screening visit: no resistance mutation to integrase inhibitors, the reverse transcriptase resistant mutations M184V plus one TAM are allowed.
* Patient enrolled in or a beneficiary of a Social Security program (State Medical Aid or AME is not a Social Security program)
* Informed consent form signed by patient and investigator

Exclusion Criteria:

* HIV-2 infection
* Currently receiving one of the following drugs: Hypericum perforatum, rifampicin, rifabutin, carbamazepine, oxcarbazepine, phenobarbital, phenytoin, sucralfate, cyclosporine, primidone, ténofovir et adéfovir.
* Hemoglobin < 10g/dL
* Platelets < 100 000/mm3
* Hepatic transaminases AST and ALT > 3x upper limit of normal (ULN)
* Severe hepatic insufficiency (Child Pugh Class C)
* Creatininemia clairance < 30 mL/min (MDRD)
* History or presence of allergy to the trial drugs or their components
* Patients participating in another clinical trial including an exclusion period that is still ongoing during the screening phase
* Patients under judicial protection due to temporarily and slightly diminished mental or physical faculties or under legal guardianship.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2020-08-17 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Virological failure is defined by plasma HIV RNA > 50 cps/mL on 2 following samples at 2 to 4 weeks apart | Week 24
  The primary outcome is the proportion of patients with virological failure at Week 24.

SECONDARY OUTCOMES:
Charlson and Fried Score | Day 1, Week 24 and Week 48
  • Assessment of co morbidities and frailty
DAD Score | Day 1,Week 24 and Week 48
  • Assessment of cardio vascular risk
polymedication | Baseline, Week 24 and Week 48
  • Assessment of polymedication and potential drug-drug interactions
drug interactions | Baseline To Week 48
  • Change of drug-drug interactions
• adverses events | Baseline To Week 48
  Rate of participants withdrawn from the study for grade 3 or 4 adverse event
therapeutic success | Week 24 and Week 48
  • Rate of therapeutic success
Viral load detectable | From Baseline to Week 48
  • Rate of participants with detectable signal in case viral load is less than 20 c/ml threshold (Cobas/TaqmanHIV-1 Roche Diagnostics) at W24 and W48
Blip detectable | Baseline to Week 48
  • Rate of participants with a blip
mutation | Day 1 to Week 48
  • Emergence of resistance mutations at time of virological failure
immunology parameters | Baseline, to Week 24 and Week 48
  • Change of CD4 and CD8 cell count from BSL,
lipid parameters | Baseline, Week 24, Week 48
  • Evolution of lipid parameters
Renal parameters | Baseline,Week 4,Week 12,Week 24 and Week 48 ;
  Renal glomerular filtration, creatinine clearance
pharmacology | Baseline, Week 12, Week 24, Week 48
  • Plasma levels of antiretroviral drugs (TAF, FTC, BIC)
Addherence | Baseline, Week 24 and Week 48
  • Adherence to treatment: self-administered questionnaire
Tolerance | Week 4, Week 24 and Week 48
  • Tolerance to treatment: questionnaire
Renal parameters (Urine) | Baseline, Week 24, Week 48
  urine albumin, urine creatinine, urine protein, beta-2-microglobulin and retinol binding protein

CONTACTS AND LOCATIONS:
Locations (8):
- France (8):
  - Hopital Sainte Marguerite, Marseille
  - Hopital Hotel Dieu, Nantes
  - Hopital L'Archet, Nice
  - Hôpital Hotel Dieu, Paris
  - Bichat Hospital, Paris
  - CH de Saint Nazaire, Saint-Nazaire
  - Hopital Gustave Dron, Tourcoing
  - Hopital Bretonneau, Tours

IPD SHARING:
Plan to Share IPD: No